CLINICAL TRIAL: NCT07263737
Title: Effectiveness of Pulsed Electromagnetic Field Therapy on Neuropathic Pain and Disability in Patients With Lumbar Disc Herniation: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Pulsed Electromagnetic Field Therapy for Neuropathic Pain in Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Gunay, MD, Medical Doctor, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2022/KK/124
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Disc Herniation With Radiculopathy
Keywords: pulsed electromagnetic field; neuropathic pain; lumbar disck herniation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed electromagnetic field (PEMF) and physical therapy (Experimental): The physical therapy protocol was arranged as follows: 20 minutes of hot pack application to the lumbar region, 10 minutes of rest, 20 minutes of conventional transcutaneus electrical nerve stimulation (TENS) applied to the lumbar region and along the radicular pain pathway, followed by another 10 minutes of rest, and finally 30 minutes of magnetic field therapy . One session lasted a total of 90 minutes.
  On the first day, patients were thoroughly instructed in a home exercise program that included lumbar isometric strengthening, pelvic tilt exercises, hamstring stretching, and core stabilization exercises. They were asked to perform each exercise twice daily with ten repetitions throughout the physical therapy program.
  Patients received one session per day, five days per week, for a total of 15 sessions.
  Interventions: Device: Pulsed electromagnetic field (PEMF)
- Sham Pulsed electromagnetic field (PEMF) and physical therapy (Sham Comparator): The physical therapy protocol was arranged as follows: 20 minutes of hot pack application to the lumbar region, 10 minutes of rest, 20 minutes of conventional transcutaneus electrical nerve stimulation (TENS) applied to the lumbar region and along the radicular pain pathway, followed by another 10 minutes of rest, and finally 30 minutes of sham magnetic field therapy . One session lasted a total of 90 minutes.
  On the first day, patients were thoroughly instructed in a home exercise program that included lumbar isometric strengthening, pelvic tilt exercises, hamstring stretching, and core stabilization exercises. They were asked to perform each exercise twice daily with ten repetitions throughout the physical therapy program.
  Patients received one session per day, five days per week, for a total of 15 sessions.
  Interventions: Device: Sham PEMF

INTERVENTIONS:
Device: Pulsed electromagnetic field (PEMF) — In our study, the device used for PEMA application was the BTL-4000 Smart. The PEMA waves applied to the treatment group were elongated square-wave signals with a frequency of 55.55 Hz and a magnetic flux density of 30 mT. A 60-cm solenoid applicator of the device was used. With this applicator, a 30-minute treatment was delivered to cover the lumbar region.
  Arms: Pulsed electromagnetic field (PEMF) and physical therapy
Device: Sham PEMF — Sham application with the same device
  Arms: Sham Pulsed electromagnetic field (PEMF) and physical therapy

SUMMARY:
This randomized controlled study evaluated whether adding pulsed electromagnetic field (PEMF) therapy to conventional physical therapy provides additional benefits for neuropathic pain and disability in patients with lumbar disc herniation (LDH).

→ This study randomly assigned patients into groups to compare treatments. It examined whether adding pulsed electromagnetic field (PEMF) therapy to standard physical therapy could give extra improvement in nerve-related pain and daily function in people with a slipped disc in the lower back.

Fifty-two patients with ≥3 months of radicular and neuropathic symptoms were enrolled and randomly assigned to a treatment group (PEMF + conventional therapy) or a control group (sham PEMF + conventional therapy).

→ Fifty-two patients who had leg pain and nerve-related symptoms for at least three months joined the study. They were randomly placed into either a treatment group (which received PEMF plus regular therapy) or a control group (which received a fake PEMF treatment plus regular therapy).

Both groups received transcutaneous electrical nerve stimulation, hot packs, and a lumbar exercise program for 15 sessions.

→ Both groups also received the same standard treatments: electrical nerve stimulation, hot packs, and a lower-back exercise program for 15 sessions.

Clinical outcomes-including Visual Analog Scale (VAS), pressure pain threshold, Modified Schober test, DN4, PainDetect, Oswestry Disability Index (ODI), and SF-36-were assessed at baseline, post-treatment, and one month after treatment.

→ Several health measures were checked before treatment, right after treatment, and again one month later. These included pain level (VAS), how sensitive the area was to pressure, lower-back flexibility, nerve-pain questionnaires (DN4 and PainDetect), disability level (ODI), and overall quality of life (SF-36).

Forty-six patients completed the study. → A total of 46 patients finished the study.

Both groups showed significant improvements in VAS scores, neuropathic pain questionnaires (DN4, PainDetect), ODI, and several SF-36 subscales (physical functioning, role-physical, and pain), with additional improvements in emotional role and social functioning observed only in the PEMF group.

→ Both groups improved in many areas: pain levels, nerve-pain scores, disability, and some parts of quality of life (such as physical functioning, daily roles, and pain). Only the PEMF group showed extra improvement in emotional well-being and social activities.

However, none of the between-group comparisons demonstrated significant differences.

* However, when the two groups were compared to each other, there were no meaningful differences.

No meaningful changes were found in lumbar flexibility or pressure pain thresholds in either group.

→ Neither group showed important changes in lower-back flexibility or in how much pressure they could tolerate on painful areas.

In conclusion, adding PEMF therapy to conventional physical therapy did not provide additional benefit for neuropathic symptoms, radicular pain, disability, lumbar flexibility, pressure pain threshold, or quality of life in patients with LDH-related neuropathic pain.

→ In summary, adding PEMF therapy to regular physical therapy did not give extra benefits for nerve pain, leg pain, disability, back flexibility, sensitivity to pressure, or quality of life in people with nerve-related pain caused by a slipped disc.

ELIGIBILITY:
Inclusion Criteria:

* • Radicular pain and neuropathic symptoms lasting longer than 3 months

  * Presence of lumbar disc herniation on lumbar MRI
  * Age between 18 and 75 years
  * Visual Analog Scale (VAS) ≥ 4
  * DN4 ≥ 4
  * At least one positive test among Straight Leg Raise Test (SLRT) and femoral stretch test
  * Patients without cognitive impairment who are able to follow verbal instructions

Exclusion Criteria:

-• Having undergone an interventional lumbar injection within the last 3 months

* Receiving physical therapy within the last 3 months
* Using medical treatment for neuropathic pain within the last 3 months
* History of lumbar surgery
* Presence of another neurological disorder that could cause neuropathic symptoms
* Cauda equina syndrome
* History of malignancy
* Uncontrolled cardiopulmonary disease
* Pregnancy
* Presence of a pacemaker or electronic implant
* Presence of diabetic neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
VAS | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  Visual Analog Scale (VAS): VAS is the most frequently used parameter for measuring pain intensity in low back pain studies. It is a self-reported scale that typically consists of a 10-cm horizontal or vertical line with two verbal descriptors placed at each end to indicate the extremes of pain. Patients are asked to mark the point that best represents their pain. The VAS score is obtained by measuring the distance in centimeters from the starting point to the patient's mark. In our study, VAS was used to assess the pain experienced by patients in the low back and leg regions during the previous week. VAS was evaluated in three different conditions: at rest, during movement, and at night.
PPT | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  Pressure Pain Threshold (PPT) Measurements with an Algometer:
  An algometer is a pressure-measuring device with a 1-cm rounded tip. The sensation of pressure and pain occurs when polymodal nociceptive nerve endings in superficial and deep tissues are stimulated. Algometers are used in clinical studies to measure the pressure pain threshold.
  After the measurement points are identified, the rounded tip of the device is placed perpendicular to the surface of the body being examined. Pressure is increased continuously at a rate of approximately 1 kg per second. Patients are instructed to indicate the moment they first feel any pain or discomfort. As soon as they report this sensation, the pressure is stopped and the pressure pain threshold value is read from the device .
  In our study, PPTmeasurements obtained with an algometer were used to evaluate the patients' pain sensitivity. The Jtech Commander Algometer was used as the device.

SECONDARY OUTCOMES:
Neuropathic pain | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  DN4 and PainDetect Questionnaire (PDQ)
Physical examination tests | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  Straight Leg Raise Test (SLRT), femoral stretch test, and the Modified Schober test
Disability | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  Oswestry Disability Index (ODI)
Quality of life Short Form-36 (SF-36) questionnaire | Patients were evaluated before treatment, at the end of treatment, and at the first month after treatment.
  The SF-36 questionnaire was developed by Ware as a general assessment tool intended for use in many diseases, evaluating quality of life through physical and mental health parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Training and Research Hospital Physical Rehabilitation and Medicine Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study data are available with the researcher and can be provided to the relevant authorities if required.